CLINICAL TRIAL: NCT02141685
Title: Correlating Time-Lapse Parameters Detected by Eeva™ With Array-Comparative Genomic Hybridization Results and Ongoing Pregnancy Rates (aCGH Study)
Brief Title: Correlating Time-Lapse Parameters With aCGH Testing in IVF Treatment (aCGH Study)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-AUX-011
Record Dates: First submitted 2014-05-13; First posted 2014-05-19 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Infertility
Keywords: in vitro fertilization; assisted reproduction techniques; noninvasive imaging of embryos; time lapse imaging of embryos; traditional morphological grading of embryos; prediction of blastocysts; infertility; preimplantation genetic diagnosis; array-Comparative Genomic Hybridization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IVF patients undergoing aCGH Testing: Women undergoing fresh IVF treatment and array-comparative genomic hybridization testing (aCGH), as recommended based on medical need by the clinical site reproductive endocrinologist.

SUMMARY:
The purpose of this research study protocol is to collect imaging data on embryos followed to blastocyst stage (Day 5-6) and correlate Eeva parameters with array - Comparative Genomic Hybridization (aCGH) results and ongoing pregnancy rates.

DETAILED DESCRIPTION:
The present study was designed to determine if there is a correlation between the Eeva System parameters and aCGH testing results. Embryos will be selected for transfer based on aCGH results and morphology. The Clinical site will have no access to the Eeva analysis at the time of the transfer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≤43 years of age.
* Women undergoing IVF treatment with planned aCGH testing using her own eggs or donor eggs.
* Antral Follicle Count ≥ 6 at time of cycle start
* Baseline (day 2-3 of cycling) FSH ≤ 15 mIU/ml
* Antimüllerian Hormone level ≥ 0.5 ng/mL
* Fertilization using only ejaculated sperm (fresh or frozen) - no surgically retrieved sperm.
* Willing to have all 2PN embryos monitored by Eeva
* Not previously enrolled in this study.
* Willing to comply with study protocol and procedures and able to speak English.
* Willing to provide written informed consent.

Exclusion Criteria:

* BMI ≥ 40
* Prior IVF cycle with < 4 x 2PN
* Planned Day 3 Assisted Hatching

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing fresh IVF treatment and undergoing aCGH testing, as recommended based on medical need by the clinical site reproductive endocrinologist.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Eeva time-lapse parameters and aCGH testing results | 5-6 days
  Analysis of correlation between time-lapse parameters collected by the Eeva System and array-Comparative Genomic Hybridization (aCGH) results

SECONDARY OUTCOMES:
Embryo Implantation Rate | 6 weeks
  Correlation of time-lapse parameters collected by Eeva and implantation rate
Clinical Pregnancy Rate | 6 weeks
  Correlation of time-lapse parameters collected by Eeva and clinical pregnancy rate
Ongoing pregnancy rate | 8-12 weeks
  Correlation of time-lapse parameters collected by Eeva and ongoing pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Shehua Shen, MD, ELD, Study Director — Progyny, Inc.
Locations (1):
- Main Line Fertility, Bryn Mawr, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.auxogyn.com